CLINICAL TRIAL: NCT01247415
Title: Clinical Investigation of Anaphylaxis, Allergic-like Reactions and Oculo-Respiratory Syndrome (ORS) Following Administration of an Adjuvanted Vaccine Against H1N1 Pandemic Influenza
Brief Title: Clinical Investigation on Allergic-like Reactions and Oculo-respiratory Syndrome After the H1N1 Pandemic Vaccine
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: PHAC/CIHR Influenza Research Network (Other Government)
Collaborators: Institut National en Santé Publique du Québec (Other); Laval University (Other); University of British Columbia (Other); Stollery Children's Hospital (Other); University of Manitoba (Other); University of Toronto (Other); CHU de Quebec-Universite Laval (Other); St. Justine's Hospital (Other); Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other); Centre hospitalier de l'Université de Montréal (CHUM) (Other); Montreal Children's Hospital of the MUHC (Other); Montreal General Hospital (Other); Hopital Charles Lemoyne (Other); IWK Health Centre (Other); Université de Montréal (Other); University of Cincinnati (Other); McMaster University (Other); Public Health Agency of Canada (PHAC) (Other Government); British Columbia Centre for Disease Control (Other Government)
Responsible Party: Principal Investigator, Gaston De Serres, Epidemiologist at the National Institute of Public Health of Quebec and professor of epidemiology at the University Laval, PHAC/CIHR Influenza Research Network
Other Study IDs: pcirn-clin-invest-aller-1011
Record Dates: First submitted 2010-11-22; First posted 2010-11-24 (Estimated); Last update posted 2012-07-04 (Estimated); Status verified 2012-07

CONDITIONS: Anaphylaxis; Allergy; Oculorespiratory Syndrome; Allergic-like Reactions
Keywords: anaphylaxis; allergy; IgE mediated; ORS; oculorespiratory syndrome; Allergic-like reactions; H1N1; Arepanrix
MeSH Terms: conditions — Anaphylaxis; Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — whole blood,PBMC and serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Anaphylaxis: Anaphylaxis: these patients will have to meet at least level 3 of diagnostic certainty according to the Brighton Collaboration criteria for anaphylaxis
- Allergic-like reactions: Allergic-like reactions: These patients will have to have displayed at least one sign or symptom of an allergic reaction (any of the minor or major criteria of anaphylaxis) but will exclude patients with conjunctivitis who will belong to the ORS group
- ORS cases: ORS cases: According to the Public Health Agency case definition, these patients should have presented a bilateral conjunctivitis plus ≥1 of the seven respiratory symptoms (cough, wheeze, chest tightness, difficulty breathing, difficulty swallowing, hoarseness or sore throat) that started within 24 hrs of vaccination, with or without facial oedema (no restriction for duration) (ref: Public Health Agency of Canada: User Guide: Report of Adverse Events Following Immunization (AEFI) Appendix III National Case Definitions of AEFIs of Special Interest: oculo-respiratory Syndrome. http://www.phac-pc.gc.ca/im/aefi_guide/ann3-eng.php
- Controls: Controls will be individuals who received the pH1N1 vaccine but did not present any of the above mentioned adverse events after their vaccine.

SUMMARY:
During the 2009-2010 immunization campaign against pandemic H1N1, some people reported having allergic-like reactions (anaphylaxis(a shock-like reaction), hives, swelling, etc.). A vaccine allergy may be more or less severe or intense. Patients may have skin reactions (rash with or without itching), respiratory problems (cough, spasm of the airways), angioedema (swelling) of various body parts (face, eyelids, throat etc.) and circulatory problems (low blood pressure or shock). Anaphylaxis is a severe allergic reaction that can sometimes be fatal. Other people vaccinated against pandemic H1N1 had an oculo-respiratory syndrome. Oculo-respiratory syndrome (ORS) is also a reaction to the influenza vaccine, which includes symptoms such as bilateral conjunctivitis (red eyes) with swelling of the face or respiratory symptoms (chest tightness, coughing, a sensation of throat closure, difficulty swallowing, hoarseness, wheezing or difficulty breathing). The investigators know that ORS is not a true allergic reaction. Because many signs and symptoms of ORS are similar to those observed during an allergic reaction, it is often difficult to distinguish ORS from an allergic reaction.

This study will compare three groups of patients: those who had allergic-like reactions, those who had ORS and vaccinated individuals who had no such adverse events. Pregnant women cannot participate in this study. The study has three goals. First, the investigators want to determine, among those who had allergic-like reactions after influenza vaccination, what proportion (percentage) of these people are actually allergic to the vaccine or its components. Second, among those who are not allergic to the vaccine, which other processes may have caused these symptoms. Finally, the investigators will try to identify whether there are features that distinguish patients who have a true allergic reaction from those affected by ORS, and those that had no adverse events.

ELIGIBILITY:
case:

Inclusion Criteria:

* There will be three groups of cases. For all groups of cases, patients will be included if the time of onset of their first symptoms has been within 24 hours after vaccination and if they are between 10 and 64 years of age.
* Anaphylaxis: these patients will have to meet at least level 3 of diagnostic certainty according to the Brighton Collaboration criteria for anaphylaxis
* Allergic-like reactions: These patients will have to have displayed at least one sign or symptom of an allergic reaction (any of the minor or major criteria of anaphylaxis) but will exclude patients with conjunctivitis who will belong to the ORS group (see below).
* ORS cases: According to the Public Health Agency case definition, these patients should have presented a bilateral conjunctivitis plus ≥1 of the seven respiratory symptoms (cough, wheeze, chest tightness, difficulty breathing, difficulty swallowing, hoarseness or sore throat) that started within 24 hrs of vaccination, with or without facial oedema (no restriction for duration)
* Controls will be individuals between 10 and 64 years of age who received the pH1N1 vaccine but did not present any of the above mentioned adverse events after their vaccine (anaphylaxis, allergic like reactions and SOR).

Exclusion Criteria:

-Pregnant women cannot participate in this study.

Ages: 10 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: During the 2009-2010 immunization campaign against pandemic H1N1, the Canada has immunized most of its population with a dose-sparing adjuvanted vaccine produced by GlaxoSmithKline (GSK). Following the vaccination, some people reported having allergic-like reactions (anaphylaxis, oculo-respiratory syndrome and allergy). This study will compare three groups of patients (cases): those who had allergic-like reactions, those who had anaphylaxis and those who had ORS post vaccination to vaccinated individuals who had no such adverse events (controls).
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2011-01; Primary Completion 2011-03 (Actual); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
proportion of individuals with IgE mediated allergic reaction | one year
  The overall objective of this clinical investigation is to estimate the proportion of individuals with IgE mediated allergic reaction to Arepanrix or its components among patients with anaphylaxis/allergic reaction after pH1N1 vaccination, and the proportion that are allergic to the 2010-2011 trivalent inactivated seasonal influenza vaccine (TIV).

SECONDARY OUTCOMES:
Biomarkers that may allow differentiation between ORS and type I hypersensitivity | two year
  We will try to identify biomarkers that may allow differentiation of patients with ORS and those with type I hypersensitivity to the vaccine.

CONTACTS AND LOCATIONS:
Locations (7):
- Canada (7):
  - Centre Hospitalier Charles Lemoyne, Greenfield Park, Quebec
  - Centre Hospitalier Universitaire de Montréal, Montreal, Quebec
  - Montreal General Hospital, Montreal, Quebec
  - Montreal Children's Hospital, Montreal, Quebec
  - Hôpitale Ste-Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Québec, Québec, Quebec
  - Centre Hospitalier et Universitaire de Sherbrooke, Sherbrooke, Quebec